CLINICAL TRIAL: NCT04653922
Title: Evaluation of Safety and Efficacy of Intrastromal Implantation of LinkCor Bioengineered Corneal Implant for Management and Treatment of Keratoconus: a Prospective, Non-randomized, Non-controlled Case Series.
Brief Title: Evaluation of Safety and Efficacy of a Bioengineered Corneal Implant for Treatment of Keratoconus
Acronym: LinkCor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LinkoCare Life Sciences AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG-PRT-001
Record Dates: First submitted 2020-11-23; First posted 2020-12-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Keratoconus
Keywords: corneal blindness; keratoconus; bioengineered cornea; intrastromal implantation; femtosecond laser
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bioengineered corneal substitute (Experimental): A cell-free, sterilized bioengineered corneal substitute made from medical grade collagen
  Interventions: Device: LinkCor Bioengineered Corneal Implant

INTERVENTIONS:
Device: LinkCor Bioengineered Corneal Implant — Intrastromal implantation of a bioengineered corneal equivalent device

SUMMARY:
This is a prospective, Phase I open-label safety study to evaluate the safety, feasibility and initial efficacy of a bioengineered corneal stromal substitute after implantation into the stroma of adults with advanced keratoconus. The bioengineered substitute and implantation technique may provide a less invasive treatment option for advanced keratoconus than current surgical approaches, that additionally does not rely on the limited availability of human donor corneal tissue.

DETAILED DESCRIPTION:
This is a Phase I, open-label, non-randomized, non-controlled ongoing clinical case series in two participating centers in Indian and Iranian hospitals, to evaluate the safety and feasibility of minimally-invasive surgery of advanced keratoconus using a bioengineered corneal stromal substitute on a compassionate basis to alleviate blindness and low vision, due to the severely limited availability of human corneal donor tissue at these centers relative to the medical need. Patients fulfilling inclusion criteria are recruited consecutively and implanted intra-stromally with the bioengineered substitute, as a less invasive surgery than full-thickness or anterior lamellar corneal transplantation. In the first phase of the study, a total of 20 patients were recruited and safety and efficacy outcomes were evaluated in those having a minimum of 12 months of postoperative follow-up. In the second phase of the study (currently ongoing), up to 40 patients are being recruited, with one-year postoperative outcomes of all included patients to be evaluated as the final study endpoint. Primary safety and efficacy outcomes will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Advanced keratoconus (according to Amsler-Krumeich classification)
* No corneal scar
* Male or female aged ≥ 18 years, no upper age limit
* Subjects indicated for a first corneal stromal transplantation (treatment naïve)
* Corneal thickness (including epithelium) at least 300µm centrally, as measured by OCT.
* Patients who gave their written signed and dated informed consent for participation

Exclusion Criteria:

* Prior corneal surgery (e.g., refractive surgery, cataract, collagen cross-linking, endothelial keratoplasty, etc.)
* Dry eye / tear film pathology
* Active ocular infection
* Glaucoma / ocular hypertension
* Active corneal ulceration
* Acute or chronic disease or illness that would increase the operation risk or confound the outcomes of the study (immune- compromised, connective tissue disease, clinically significant atopic disease, etc.)
* Any other medical condition that in the judgment of the clinical investigator or corneal surgeon is not compatible with the study procedures
* General history judged by the investigator to be incompatible with the study (e.g., life-threatening patient condition, other condition where postoperative follow-up may be difficult).
* known diabetes or other neuro-degenerative disorder (as corneal nerves can be affected leading to impaired wound healing)
* Inability of patient to understand the study procedures and thus inability to give informed consent.
* Participation in another clinical study within the last 3 months
* Already included once in this study (can only be included for one treated eye).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Safety outcome measure | 6 months
  The primary safety endpoint is defined such that a rejection leading to implant removal should occur in no more than 10% of implanted eyes. The implant rejection is defined as a clinical situation when the implanted eye has decreased central corneal clarity and decreased implant clarity, corneal vascularization inside of laser created pocket and inflammation.
Corneal curvature measured by keratometry (efficacy measure) | 6 months
  The maximum and minimum corneal curvature (steepness) of each eye will be measured by a keratometer and reported in diopter (D) unit and represented as "K-value". The efficacy outcome is that more than 60% of the eyes should have a decrease in K-value at 6 months postoperatively.
Central corneal thickness measured by topography techniques (efficacy measure) | 6 months
  Central corneal thickness (CCT) will be measured in microns and reported using a two-dimensional thickness map made by optical coherence tomography (OCT) and/or Pentacam topography. The efficacy outcome is that more than 60% of the eyes should have an increase in CCT at 6 months postoperatively.
Visual acuity (efficacy measure) | 6 months
  Vision improvement equivalent of minimum one line in Snellen chart in uncorrected distance visual acuity (UDVA) or corrected distance visual acuity (CDVA).

CONTACTS AND LOCATIONS:
Overall Officials: Namrata Sharma, MD, Principal Investigator — ALL INDIA INSTITUTE OF MEDICAL SCIENCES, Dr. R. P. Centre for Ophthalmic Sciences, AIIMS, New Delhi; Mahmoud Jabbarvand Behrouz, MD, Principal Investigator — University of Tehran, Farabi Eye Hospital
Locations (2):
- All India Institute of Medical Sciences, Dr. R. P. Centre for Ophthalmic Sciences, AIIMS,, New Delhi, India
- Farabi Eye Hospital, Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rafat M, Jabbarvand M, Sharma N, Xeroudaki M, Tabe S, Omrani R, Thangavelu M, Mukwaya A, Fagerholm P, Lennikov A, Askarizadeh F, Lagali N. Bioengineered corneal tissue for minimally invasive vision restoration in advanced keratoconus in two clinical cohorts. Nat Biotechnol. 2023 Jan;41(1):70-81. doi: 10.1038/s41587-022-01408-w. Epub 2022 Aug 11. PMID 35953672